CLINICAL TRIAL: NCT02309918
Title: Interferon-free Treatment of Acute Genotype 1 Hepatitis C Virus Infection With Ledipasvir/Sofosbuvir Fixed-Dose Combination - The HepNet Acute HCV IV Study
Brief Title: HepNet Acute HCV IV - LDV/SOF FDC in Acute Genotype 1 Hepatitis C Virus Infection
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: HepNet Study House, German Liverfoundation (Network)
Collaborators: Hannover Medical School (Other); Gilead Sciences (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: HepNet-aHCV-IV; 2013-001081-42 (EudraCT Number)
Record Dates: First submitted 2014-11-04; First posted 2014-12-05 (Estimated); Last update posted 2017-08-28 (Actual); Status verified 2017-08

CONDITIONS: Acute Hepatitis C
Keywords: acute HCV Genotype 1 Infection; HCV RNA; LDV/SOF FDC

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- LDV/SOF FDC (Other): Ledipasvir/Sofosbuvir fixed dose combination (FDC) tablet (LDV 90 mg/SOF 400 mg) once daily
  Interventions: Drug: LDV/SOF FDC

INTERVENTIONS:
Drug: LDV/SOF FDC — Ledipasvir/Sofosbuvir fixed dose combination (FDC) tablet (LDV 90 mg/SOF 400 mg) once daily

SUMMARY:
This is an open-label, single arm, multicenter, pilot-study to compare the efficacy and safety of LDV/SOF fixed dose combination (FDC) in subjects with acute genotype 1 HCV infection. A total of 20 subjects will be assigned to receive LDV/SOF FDC tablet (LDV 90 mg/SOF 400 mg/) once daily for 6 weeks.Patients will be followed up for 24 weeks.

ELIGIBILITY:
Inclusion Criteria:

1. Willing and able to provide written informed consent
2. Male or female, age ≥ 18 years
3. HCV RNA ≥ 103 IU/mL at Screening
4. Confirmation of acute genotype 1 HCV infection documented by either:

   documented seroconversion to HCV antibody positivity within the 4 months preceding screening or known or suspected exposure to HCV within the 4 months preceding screening with 10 times elevated serum ALT Level at screening or 4 weeks preceding screening without evidence of confounding liver disorders
5. If the patient visits a physician due to symptoms of acute HCV, no greater than a 12 week interval may have elapsed between the time of the visit and screening
6. Non-cirrhotic. Absence of cirrhosis will be determined based on clinical parameters or ultrasound
7. Body mass index (BMI) ≥ 18 kg/m2
8. Screening ECG without clinically significant abnormalities
9. Subjects must have the following laboratory parameters at screening:

   1. Hemoglobin ≥ 10 g/dL
   2. Platelets ≥ 90,000/µL
   3. INR ≤1.5 x ULN unless subject has known hemophilia or is stable on an anticoagulant regimen affecting INR
   4. Albumin ≥ 3 g/dL
   5. HbA1c ≤ 10%
   6. Creatinine clearance (CLcr) ≥ 60 mL/min, as calculated by the Cockcroft- Gault equation
10. Subject has not been treated with any investigational drug or device within 42 days of the Screening visit
11. A negative serum pregnancy test is required for female subjects (unless surgically sterile or women ≥ 54 years of age with cessation for 24 ≥ months of previously occurring menses).

    Complete abstinence from intercourse. Periodic abstinence (e.g., calendar, ovulation, symptothermal, post-ovulation methods) is not permitted.

    Or

    Consistent and correct use of 1 of the following methods of birth control listed below, in addition to a male partner who correctly uses a condom, from the date of Screening until 30 days after last dose of study drug:
    * intrauterine device (IUD) with a failure rate of < 1% per year
    * female barrier method: cervical cap or diaphragm with spermicidal agent
    * tubal sterilization
    * vasectomy in male partner
    * hormone-containing contraceptive:
    * implants of levonorgestrel
    * injectable progesterone
    * oral contraceptives (either combined or progesterone only)
    * contraceptive vaginal ring
    * transdermal contraceptive patch
12. Male subjects must agree to refrain from sperm donation from the day of screening and for at least 90 days after the last dose of study drug.
13. Subject must be of generally good health as determined by the Investigator.
14. Subject must be able to comply with the dosing instructions for study drug administration and be able to complete the study schedule of assessments.

Exclusion Criteria:

1. Clinically-significant illness (other than HCV) or any other major medical disorder that, in the opinion of the investigator, may interfere with subject treatment, assessment or compliance with the protocol; subjects currently under evaluation for a potentially clinically-significant illness (other than HCV) are also excluded.
2. Gastrointestinal disorder or post operative condition that could interfere with the absorption of the study drug (for example, gastric bypass or severe ulcerative colitis).
3. Difficulty with blood collection and/or poor venous access for the purposes of phlebotomy.
4. Clinical hepatic decompensation (i.e., clinical ascites, encephalopathy or variceal hemorrhage).
5. Solid organ transplantation.
6. Significant pulmonary disease or significant cardiac disease.
7. Psychiatric hospitalization, suicide attempt, and/or a period of disability as a result of their psychiatric illness within the last 2 years. Subjects with psychiatric illness that is well-controlled on a stable treatment regimen for at least 12 months prior to screening or has not required medication in the last 12 months may be included.
8. Malignancy within 5 years prior to screening, with the exception of specific cancers that are entirely cured by surgical resection (basal cell skin cancer, etc). Subjects under evaluation for possible malignancy are not eligible.
9. Significant drug allergy (such as anaphylaxis or hepatotoxicity).
10. Any prior treatment for HCV infection including prior exposure to any inhibitor of the NS5B and NS5A.
11. Pregnant or nursing female or male with pregnant female partner
12. Chronic liver disease of a non-HCV etiology (e.g., hemochromatosis, autoimmune hepatitis, alcoholic liver disease, Wilson's disease, α1 antitrypsin deficiency, cholangitis)
13. Infection with hepatitis B virus (HBV; defined as HBsAg-positive) or human immunodeficiency virus (HIV)
14. Chronic use of systemically administered immunosuppressive agents (e.g., prednisone equivalent > 10 mg/day)
15. Clinically-relevant drug or alcohol abuse within 12 months of screening including any uncontrolled drug use within 6 months of screening. A positive drug screen will exclude subjects unless it can be explained by a prescribed medication; the diagnosis and prescription must be approved by the investigator. Uncontrolled users of intravenous drugs will not be permitted to enroll in the study.
16. Donation or loss of more than 400 ml blood within 2 months prior to Baseline/Day 1
17. Use of any prohibited concomitant medications within 21 days of the Baseline/Day 1 visit, this washout period does not apply to proton pump inhibitors, which can be taken up to 7 days before Day 1.
18. Known hypersensitivity to LDV, SOF or formulation excipients

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2014-11; Primary Completion 2016-08 (Actual); Study Completion 2016-08 (Actual)

PRIMARY OUTCOMES:
Efficacy of treatment with ledipasvir (LDV)/sofosbuvir (SOF) FDC (proportion of subjects with sustained viral response (HCV RNA < LLOQ TND) using COBAS TaqMan Realtime PCR) | 12 weeks
  To evaluate the efficacy of treatment with ledipasvir (LDV)/sofosbuvir (SOF) FDC for 6 weeks in patients with acute genotype 1 HCV infection as measured by the proportion of subjects with sustained viral response (HCV RNA < LLOQ TND) 12 weeks after discontinuation of therapy (SVR 12) using COBAS TaqMan Realtime PCR.
Safety and tolerability of LDV/SOF FDC-containing regimens (frequency of AEs and SAEs) | 24 weeks after treatment
  To evaluate the safety and tolerability of LDV/SOF FDC-containing regimens administered for up to 6 weeks in patients with acute genotype 1 HCV infection as measured by the frequency of AEs and SAEs assessed at end of treatment, 12 and 24 weeks after end of treatment.

SECONDARY OUTCOMES:
Durability of response (proportion of subjects with sustained viral response (HCV RNA < LLOQ TND) | 24 weeks after treatment
  To determine the durability of response after discontinuation of therapy as measured by the proportion of subjects with sustained viral response (HCV RNA < LLOQ TND) 24 weeks after discontinuation of therapy (SVR 24).
Kinetics of circulating HCV RNA (mean viral load) | 24 weeks after treatment
  To evaluate the kinetics of circulating HCV RNA measured as mean viral load during treatment (Baseline, week 2,4,6) and after treatment discontinuation (Follow up week 4, 12, 24)
Emergence of viral resistance to LDV/SOF FDC | 24 weeks after treatment
  To evaluate the emergence of viral resistance to LDV/SOF FDC during treatment and after treatment discontinuation

OTHER OUTCOMES:
HCV-specific T cell responses | 24 weeks after treatment
  To assess any relationship between HCV-specific T cell responses and treatment efficacy
Relationship between NK cell phenotype and function and treatment efficacy | 24 weeks after treatment
  To assess any relationship between NK cell phenotype and function and treatment efficacy
Relationship between circulating serum chemokines and treatment efficacy and safety | 24 weeks after treatment
  To assess any relationship between circulating serum chemokines and treatment efficacy and safety

CONTACTS AND LOCATIONS:
Overall Officials: Michael P. Manns, Prof. Dr., Principal Investigator — MHH, Klinik für Gastroenterologie, Hepatologie und Endokrinologie, Carl-Neuberg-Str. 1, 30625 Hannover, Germany
Locations (20):
- Germany (20):
  - • Charite, Universitätsmedizin Berlin, Campus Virchow-Klinikum, Medizinische Klinik mit Schwerpunkt Hepatologie und Gastroenterologie, Berlin
  - Universitätsklinikum Bonn, Medizinische Klinik und Poliklinik I, Bonn
  - Medizinisches Versorgungszentrum, Düsseldorf
  - • Universitätsklinikum Essen, Klinik für Gastroenterologie und Hepatologie, Essen
  - Universitätsklinikum Frankfurt, Medizinische Klinik 1, Frankfurt
  - Universitätsklinikum Freiburg, Klinik für Innere Medizin II, Gastroenterologie, Hepatologie, Endokrinologie und Infektiologie, Freiburg im Breisgau
  - Ifi, Institut für Interdisziplinäre Medizin, Hamburg
  - Universitätsklinikum Hamburg-Eppendorf, Medizinische Klinik und Poliklinik, Hamburg
  - Medizinische Hochschule Hannover, Klinik für Gastroenterologie, Hepatologie und Endokrinologie, Hanover
  - Universitätsklinikum Heidelberg, Gastroenterologie, Infektionen, Vergiftungen, Heidelberg
  - Gastroenterologische Gemeinschaftspraxis Herne, Herne
  - Universitätsklinikum des Saarlandes und Medizinische Fakultät der Universität des Saarlandes, Klinik für Innere Medizin II - Gastroenterologie und Endokrinologie, Homburg
  - Universitätsklinikum Schleswig-Holstein, Klinik für Innere Medizin 1, Gastroenterologie, Hepatologie, Ernährungs- und Altersmedizin, Kiel
  - Universitätsklinikum Leipzig, Klinik und Poliklinik für Gastroenterologie und Rheumatologie, Leipzig
  - Universitätsmedizin der Johannes Gutenberg-Universität Mainz, I. Medizinische Klinik und Poliklinik, Mainz
  - Oberberg City München, München
  - Klinikum rechts der Isar der TU-München, II. Medizinische Klinik und Poliklinik (Gastroenterologie), München
  - Medizinisches Versorgungszentrum Offenburg GmbH, St. Josefklinik, Ambulante Gastroenterologie, Offenburg
  - Universitätsklinikum Tübingen, Innere Medizin I, Hepatologie, Gastroenterologie, Infektiologie, Tübingen
  - Universitätsklinikum Würzburg,Medizinische Klinik und Poliklinik II, Zentrum Innere Medizin, Würzburg

REFERENCES:
- [Result] Deterding K, Spinner CD, Schott E, Welzel TM, Gerken G, Klinker H, Spengler U, Wiegand J, Schulze Zur Wiesch J, Pathil A, Cornberg M, Umgelter A, Zollner C, Zeuzem S, Papkalla A, Weber K, Hardtke S, von der Leyen H, Koch A, von Witzendorff D, Manns MP, Wedemeyer H; HepNet Acute HCV IV Study Group. Ledipasvir plus sofosbuvir fixed-dose combination for 6 weeks in patients with acute hepatitis C virus genotype 1 monoinfection (HepNet Acute HCV IV): an open-label, single-arm, phase 2 study. Lancet Infect Dis. 2017 Feb;17(2):215-222. doi: 10.1016/S1473-3099(16)30408-X. Epub 2016 Oct 28. PMID 28029529